CLINICAL TRIAL: NCT03701542
Title: The Application of M-charts and Microperimetry for the Assessment of Visual Function in Patients After Vitrectomy Due to the Full Thickness Macular Hole.
Status: Completed | Type: Observational
Sponsor: Medical University of Lublin (Other)
Responsible Party: Sponsor
Other Study IDs: 0003
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Macular Holes; Microperymetry; Vitrectomy; M-charts
Keywords: macular hole; microperymetry; vitrectomy; m-charts; metamorphopsia
MeSH Terms: conditions — Retinal Perforations; Vision Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group of 22 patients: Group of 22 patients who underwent vitrectomy due to macular hole
  Interventions: Diagnostic Test: Microperymetry; Diagnostic Test: M-charts

INTERVENTIONS:
Diagnostic Test: Microperymetry — Microperimetry is a procedure to assess retinal sensitivity while fundus is directly examined; it enables exact correlation between macular pathology and corresponding functional abnormality.
Diagnostic Test: M-charts — The M-chart (Inami Co., Tokyo, Japan) is a diagnostic tool developed by Matsumoto to quantify the degree of metamorphopsia in patients with macular diseases.

SUMMARY:
To examine the relationship between morphological and functional results in eyes after vitrectomy due to the full thickness macular hole (FTMH).

ELIGIBILITY:
Inclusion Criteria:

The diagnosed full thickness macular hole and psuedophakia.

Exclusion Criteria:

macular pseudohole, non-full thickness macular hole, retinal detachment, other ocular comorbidities.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: 22 patients
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
The best-corrected visual acuity (BCVA) | 1 to 6 months
  Acuity is a measure of visual performance. The eye exam seeks to find the prescription that will provide the best corrected visual performance achievable
Amsler test | 1 to 6 months
  The Amsler grid, consisting of evenly spaced horizontal and vertical lines, has been widely used since 1947 to test the metamorphopsia.
Central retinal thickness | 1 to 6 months
  Quantitative thickness measurements derived from the "fast macular scan" algorithm report retinal thickness at several locations including the center point, central subfield, and 4 inner and 4 outer zones of the macula.

SECONDARY OUTCOMES:
Retinal sensitivity | 1 to 6 months
  Microperimetry is a procedure to assess retinal sensitivity while fundus is directly examined; it enables exact correlation between macular pathology and corresponding functional abnormality. It is a psychophysical method which is rapid, safe and non-invasive.

IPD SHARING:
Plan to Share IPD: Yes
All data will be available in brief.

REFERENCES:
- [Derived] Wrzesinska D, Nowomiejska K, Nowakowska D, Toro MD, Bonfiglio V, Reibaldi M, Avitabile T, Rejdak R. Secondary Vitrectomy with Internal Limiting Membrane Plug due to Persistent Full-Thickness Macular Hole OCT-Angiography and Microperimetry Features: Case Series. J Ophthalmol. 2020 Sep 21;2020:2650873. doi: 10.1155/2020/2650873. eCollection 2020. PMID 33029387
- [Derived] Wrzesinska D, Nowomiejska K, Nowakowska D, Brzozowska A, Avitabile T, Reibaldi M, Rejdak R, Toro M. Vertical and Horizontal M-Charts and Microperimetry for Assessment of the Visual Function in Patients after Vitrectomy with ILM Peeling due to Stage 4 Macular Hole. J Ophthalmol. 2019 May 6;2019:4975973. doi: 10.1155/2019/4975973. eCollection 2019. PMID 31198606